CLINICAL TRIAL: NCT05601375
Title: Comparison of Prenatal and Postnatal Cardiac Function Assessed by Echocardiography Between Foetuses/Neonates With a Structural Heart Disease, With an Fetal Growth Restriction (FGR) and Healthy Fetuses/Neonates
Brief Title: Speckle Tracking Echocardiography in Infants, Prenatally and Postnatally
Acronym: STIPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Jerome Cornette, Dr., Erasmus Medical Center
Other Study IDs: NL80033.078.21/STIPP-study
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Speckle Tracking; Fetus Fetus; Neonate; Structural Heart Disease; Fetal Growth Restriction
MeSH Terms: conditions — Fetus-in-Fetu; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnancy with a healthy fetus: 3 times echocardiography in pregnancy once echocardiography after birth
  Interventions: Other: Echocardiography
- Pregnancy with a fetus with a structural heart disease: 3 times echocardiography in pregnancy once echocardiography after birth
  Interventions: Other: Echocardiography
- Pregnancy with a fetus with a fetal growth restriction: 3 times echocardiography in pregnancy once echocardiography after birth
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — Fetal echocardiography (ultrasound)

SUMMARY:
Comparison of prenatal and postnatal cardiac function assessed by echocardiography using pulsed wave Doppler, Tissue Doppler and speckle tracking (strain and strain rate) between foetuses/neonates with a structural heart disease, with an fetal growth restriction (FGR) and healthy fetuses/neonates.

DETAILED DESCRIPTION:
Rationale:

Currently, fetal echocardiography mainly focusses on the detection of structural heart disease. New echocardiographic techniques also permit detailed assessment of the myocardial contraction and relaxation, permitting early detection of subtle changes in heart function. Structural heart disease and fetal growth restriction are often accompanied by changes in myocardial function. These changes already start during early intrauterine life. They can influence clinical course and outcome during fetal adaptation to hypoxic intrauterine conditions, during transition from fetal to neonatal circulation and during early neonatal life in both growth restricted infants and infants with heart disease. With improved survival of these infants, it becomes clear that these changes in cardiac function, subtle in early life, often progress or induce remodelling affecting long term cardiovascular outcome. Expanding the ultrasonic examination of the heart by adding measurements related to fetal cardiac function would increase knowledge about the physiology and pathophysiology of cardiac adaptation during fetal and early neonatal life in healthy infants as well in infants with fetal growth restriction and/or a structural heart disease. Early detection of dysfunction could lead to targeted preventive strategies to improve short term and long term cardiovascular outcomes in these vulnerable children.

Early changes before overt cardiac dysfunction can be observed by analysing myocardial deformation during contraction and relaxation with ultrasonic techniques such as speckletracking (focussing on myocardial strain and strain rate) and Tissue Doppler. These techniques are validated in the adult and pediatric populations but remain experimental in fetuses. The fetal heart is much smaller, beats faster and is more difficult to assess through the maternal abdomen. Besides that, the circulation and balance between left and right ventricle is fundamentally different in a fetus. This brings challenges in technical feasibility as well as in clinical interpretation of differences. Recent technical innovations permit to overcome the former and gain experience with the latter.

Along with 2-D, 3-D and pulsed waved Doppler assessments, inclusion of these techniques could be of additional value in the assessment of the fetal heart.

Objective: Comparison cardiac function assessed by echocardiography using 2-D, 3-D, pulsed wave Doppler, Tissue Doppler and speckle tracking (strain and strain rate) between fetuses/neonates with structural heart disease, fetuses/neonates with fetal growth restriction (FGR) and healthy fetuses/neonates, both prenatally and postnatally.

Study design: A longitudinal prospective cohort study, conducted at the Department of Obstetrics and Gynaecology (Division of Fetal Medicine) and the Department of Paediatrics (Division of Paediatric Cardiology and Division of Neonatology) of the Erasmus Medical Centre Rotterdam.

Study population: Women, aged ≥16 years, with a singleton pregnancy with either a healthy fetus, a fetus with an fetal growth restriction or a fetus with structural heart disease.

Main study parameters/endpoints:

Comparison of fetal systolic and diastolic function in fetuses with a structural heart disease, fetuses with an FGR and healthy fetuses, using speckle tracking, pulsed waved Doppler and tissue Doppler, at multiple time points in the pregnancy and within 72 hours postpartum.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Burden associated with participation exists for the group with healthy fetuses of two (additional) prenatal investigations and one (additional) postnatal investigation. For the group with fetuses with a structural heart disease the burden exists of one (additional) prenatal investigation and for the group of fetuses with a growth restriction, the burden exists of one (additional) postnatal investigation. All investigations have an estimated time of 15-30 minutes. Ultrasound can be safely used in pregnancy (Doppler ultrasound can be safely used from 11 weeks in pregnancy). There is no risk associated with participation for mother and fetus. There is no individual benefit for participants.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Sufficient command of the Dutch language
* A pregnancy with a fetus with a structural heart disease, or
* A pregnancy with a fetus with an FGR (defined as: weight and/or abdominal circumference p<10, or deviating growth (weight and/or abdominal circumference) > 20 percentiles, and Doppler abnormalities in either the umbilical artery, the uterine artery or the medial cerebral artery), or
* A pregnancy with a healthy fetus (without any major fetal congenital abnormality)

Exclusion Criteria:

* Multiple pregnancy
* A pregnancy with known fetal genetic abnormality
* A pregnancy with other major fetal congenital abnormalities

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women, aged ≥16 years, with a singleton pregnancy with either a healthy fetus, a fetus with fetal growth restriction (defined as: weight and/or abdominal circumference p<10, or deviating growth (weight and/or abdominal circumference) > 20 percentiles, and Doppler abnormalities in either the umbilical artery, the uterine artery or the medial cerebral artery) or a fetus with a structural heart disease.
Sampling Method: Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2025-09-12 (Estimated); Study Completion 2025-09-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of fetal systolic and diastolic function (strain and strain rate) | 3 years

SECONDARY OUTCOMES:
Technical feasibility of cardiac function measurements of fetal echocardiography using speckle tracking, pulsed waved Doppler and Tissue Doppler in fetuses with a structural heart disease. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided